CLINICAL TRIAL: NCT06502080
Title: Standard-of-care Systemic Therapy With or Without Consolidative Radiotherapy in Patients With Oligometastatic/Locally Advanced Unresectable Biliary Tract Cancer: an Open-label, Randomised, Controlled Study
Brief Title: Consolidative Radiotherapy (CSRT) in Patients With Oligometastatic/Locally Advanced Unresectable Bilary Tract Cancer (BTC)
Acronym: RADITOP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024139; ZSLCYJ202308 (Other Grant/Funding Number: Zhongshan Hospital, Fudan University)
Record Dates: First submitted 2024-07-07; First posted 2024-07-15 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Biliary Tract Cancer
Keywords: biliary tract cancer; consolidative radiotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Cisplatin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: consolidative radiotherapy group (Experimental): patients treated with standard-of-care systemic therapy combined with consolidative radiotherapy
  Interventions: Radiation: Consolidative radiotherapy; Drug: Standard-of-care systemic therapy: Gemcitabine + cisplatin/oxaliplatin + Durvalumab/Pembrolizumab/Sintilimab/Toripalimab
- control group: standard-of-care systemic therapy alone (Other): patients treated with standard-of-care systemic therapy
  Interventions: Drug: Standard-of-care systemic therapy: Gemcitabine + cisplatin/oxaliplatin + Durvalumab/Pembrolizumab/Sintilimab/Toripalimab

INTERVENTIONS:
Radiation: Consolidative radiotherapy — Consolidative radiotherapy: total dose and number of fractions will depend on the site of disease. Treatment will be given daily, or every other day, over 1 -3 weeks. Physicians should try to give the highest BED whenever possible while respecting normal tissue tolerance. All lesions are recommended to receive a biologically effective dose (BED) of 60 Gy or higher (BED10≥70), assuming α/β ratio of 10 and using the linear-quadratic model: BED = nd x [1 + d/(α/β)] where n is number of fractions and d is dose per fraction. Sometimes BED ≥80 Gy is preferred, with lower doses ≥50 Gy allowed at the discretion of the treating physician for concerns about normal tissue toxicity.
  Arms: Experimental group: consolidative radiotherapy group
Drug: Standard-of-care systemic therapy: Gemcitabine + cisplatin/oxaliplatin + Durvalumab/Pembrolizumab/Sintilimab/Toripalimab — Standard-of-care systemic therapy as decided by the treating medical oncologist: Gemcitabine + cisplatin/oxaliplatin + Durvalumab/Pembrolizumab/Sintilimab/Toripalimab

SUMMARY:
The purpose of this clinical trial is to investigate whether the inclusion of radiotherapy, in addition to standard-of-care systemic therapy, could improve the treatment effectiveness of patients with oligometastatic/locally advanced unresectable biliary tract cancer. The primary question that the trial aims to address is: does the addition of consolidative radiotherapy to standard-of-care systemic therapy for treating oligometastatic/locally advanced unresectable biliary tract cancer, result in a prolonged progression-free survival (PFS)?

Researchers will assess whether radiotherapy can enhance PFS by comparing the survival time of patients with oligometastatic/locally advanced unresectable biliary tract cancer who receive standard-of-care systemic therapy alone versus those who receive standard-of-care systemic therapy along with consolidative radiotherapy.

Participants in this trial will:

Either receive or not receive consolidative radiotherapy following six cycles of standard-of-care systemic therapy.

DETAILED DESCRIPTION:
Standard-of-care systemic therapy with or without consolidative radiotherapy in patients with oligometastatic/locally advanced unresectable biliary tract cancer: an open-label, randomised, controlled study.

Eligible patients will be randomized in a 1:1 ratio to receive either current standard systemic therapy alone (control arm) or standard systemic therapy plus consolidative radiotherapy to all sites of known disease (experimental arm). Patients in both arms have the option of receiving upfront or subsequent standard palliative radiotherapy to any symptomatic sites requiring prompt intervention.

Because of the different treatment modalities in the study, it is not possible to blind the patient or physician to the treatment arm. Follow-ups for tumor assessment will conclude 2 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. The disease has not progressed following the restaging imaging evaluation in patients with oligometastatic/locally advanced unresectable BTC after four cycles of first-line systemic treatment.
2. Definition of oligometastatic/locally advanced unresectable BTC disease: not a candidate for surgical resection at all sites: surgery to all sites not recommended by multidisciplinary team, or unfit or declining surgery.
3. Definition of oligometastatic disease: patients with distant organ metastasis or nonregional lymph node metastasis, or distant organ/nonregional lymph node metastasis and regional lymph node metastasis, as defined by the American Joint Committee on Cancer, 8th edition. The total number of metastases is ≤5 and the number of metastases in any single organ system (e.g., lung, liver) is ≤3.
4. All sites of disease must be amenable to radiotherapy and can be safely treated. Each lesion is counted separately at the time of registration and contributes to the total number of metastases. For regional lymph nodes metastases, all positive regional lymph nodes are counted together as one lesion. For nonregional lymph node metastases, adjacent metastatic lymph nodes can be treated as one lesion. Lesions that have subsided during previous treatment (i.e., are no longer visible on CT scan or have eliminated affinity on positron emission tomography [PET]-CT) are not included in the total number. At least one metastatic lesion meets the RECIST v1.1 criteria for assessable lesions. Bone metastases without soft tissue involvement can be included but are not considered assessable lesions. However, if bone metastases have soft tissue involvement and meet the criteria for assessable lesions, they are considered measurable lesions.
5. Patients who experience recurrence after curative surgery with a time interval of >6 months can be eligible for inclusion. If adjuvant therapy (excluding radiotherapy) is administered, the patient must have completed adjuvant therapy for a period of at least 6 months before meeting the inclusion criteria.
6. Primary tumor lesions and all metastases of current diagnosis have not received local treatment, such as radiotherapy, surgery or radiofrequency ablation, prior to enrollment.
7. The patient is over 18 years old and has an Eastern Cooperative Oncology Group score of 0-1;
8. Life expectancy is greater than 12 weeks.
9. Vital organ function meets the following requirements: absolute neutrophil count ≥1.5 × 109/l; platelet count ≥100 × 109/l; hemoglobin ≥9 g/dl; serum albumin ≥2.8 g/dl; total bilirubin ≤1.5 × upper limit of normal (ULN) and alanine transaminase, aspartate aminotransferase and/or alkaline phosphatase ≤2.5 × ULN (if there is liver metastasis, alanine transaminase and/or aspartate aminotransferase ≤5 × ULN; if there is liver metastasis or bone metastasis, alkaline phosphatase ≤5 × ULN); serum creatinine ≤1.5 × ULN or creatinine clearance >60 ml/min. For patients with pulmonary lesions or previous lung irradiation who are known or suspected to have impaired lung function, the forced expiratory volume for 1 second of lung function must be above 1 l.
10. Female subjects of childbearing age must have a negative urine or serum pregnancy test within 72 h prior to randomization. Subjects must agree to adequate contraception during the trial.
11. Each patient is voluntarily enrolled, and the informed consent form is signed by the patient or their legal representative.

Exclusion Criteria:

1. Histology includes components of mixed hepatocellular carcinoma, fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, or biliary adenocarcinoma.
2. Complete response to four cycles of first-line systemic treatment (i.e. no measurable target for radiotherapy).
3. There is new metastasis during the four cycles of first-line systemic treatment and the number of metastases is more than five.
4. Patient has uncontrolled brain metastases or vertebral body metastasis with spinal cord compression symptoms.
5. The toxicity of previous antitumor treatment has not recovered to ≤1 based on National Cancer Institute Common Terminology Criteria for Adverse Events v4.03 (except for hair loss) or the level specified by the inclusion/exclusion criteria.
6. Patient has uncontrolled pleural, pericardial or pelvic effusion that requires repeated drainage.
7. Patient is a pregnant or breastfeeding woman.
8. Patient has a history of immunodeficiency or severe medical disease that is not well controlled and may have an effect on study treatment.
9. Any other malignant tumor has been diagnosed within 5 years prior to or after the diagnosis of BTC, except for malignant tumors with a low risk of metastasis and death (5-year survival rate >90%), such as well-treated basal cell or squamous cell skin cancer or cervical cancer in situ.
10. Any other condition which in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Upto 2 years
  Progression free survival is defined as the duration between the date of randomization to the date of first documented progression or death due to any cause or date of last follow-up, whichever is earlier.

SECONDARY OUTCOMES:
Overall survival (OS) | Upto 2 years
  Overall survival is defined as the duration between the date of randomization to the date of death due to any cause or the date of last follow-up, whichever is earlier.
Local control rates of treated sites | Upto 2 years
  Local control rate will be defined as the absence of progressive disease at the treated sites.
New distant metastases | Upto 2 years
  Time to onset of new distant metastases.
Response rates | From randomization every 3 months upto 2 years
  To compare response rates between the two arms.
Health Related QOL using the EORTC-QLQ-C30 questionnaire | From randomization every 3 months till 2 years
  To evaluate patient reported outcomes between the two arms. EORTC QLQ-C30 scales: global health/QoL, functional domains (physical, role, cognitive, emotional, social), and symptom scales/items (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea). Recall period: past week; response range: not at all to very much, global/QOL range: very poor to excellent. Scale score range: 0 to 100. Higher functional/global QoL score = better functioning and higher symptom score = greater degree of symptoms.
Health Related QOL using the EORTC QLQ-BIL21 questionnaire | From randomization every 3 months till 2 years
  To evaluate patient reported outcomes between the two arms. EORTC QLQ-BIL21 (European Organisation for Research and Treatment of Cancer questionnaire for measuring quality of life in patients with cholangiocarcinoma and cancer of the gallbladder), scores range from 0 to 100, where a lower score means a better quality of life.
Radiotherapy related toxicity using CTC v5.0 (radiotherapy related acute and late toxicity) | Upto 2 years
  At baseline and at subsequent follow up till 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaochong Zeng, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers in order to protect patients' privacy.